CLINICAL TRIAL: NCT05210881
Title: Weaning From Nasal High Flow Therapy: an Explorative Study Assessing the Usefulness of the ROX Index to Predict Outcome of the Weaning Process in Combination With a Withdrawal Trial
Brief Title: Weaning From Nasal High Flow Therapy
Status: Completed | Type: Observational
Sponsor: Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Professor of Intensive Care Medicine, Head of ICU, Hôpital Louis Mourier
Other Study IDs: HLM_JDR11
Record Dates: First submitted 2022-01-11; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Distress Syndrome, Adult; Acute Hypoxemic Respiratory Failure; Acute Respiratory Distress Syndrome; Weaning Failure
Keywords: nasal high flow oxygen; withdrawal from nasal high flow therapy; ROX index; acute hypoxemic respiratory failure; withdrawal trial
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nasal high flow is widely used in critically ill patients admitted to the intensive care unit (ICU) for acute hypoxemic respiratory failure. It has been shown to improve patient comfort, increase oxygenation and reduce need for intubation in some patients. The Respiratory Oxygenation (ROX) index has been established as a simple tool to help clinicians identify those patients who will succeed and those who will fail under nasal high flow and therefore predict the need for intubation. However, when nasal high flow therapy is successful, little is known as to how and when weaning of this device should be performed and what are the predictors of a safe withdrawal of the device. The objectives of this retrospective exploratory study are to identify a cut-off value of the ROX index predictive of success of the withdrawal trial, to describe a one-year use of the withdrawal trial; to describe the ROX value closest to weaning from nasal high flow, and to identify factors associated with success or failure of the withdrawal trial from nasal high flow therapy in patients receiving nasal high flow therapy.

DETAILED DESCRIPTION:
Although nasal high flow is widely used in critically ill patients admitted to the intensive care unit (ICU) for acute hypoxemic respiratory failure, and its benefits have been shown in multiple studies, little is known as to how and when weaning from the technique device should be performed and what are the predictors of a safe withdrawal. The Respiratory Oxygenation (ROX) index was established and tested to predict outcome of nasal high flow therapy in patients with acute hypoxemic respiratory failure. It combines three parameters available at the bedside that reflect patient's respiratory status: respiratory rate, the level of the inspired fraction of oxygen (FiO2) and pulse oximetry (SpO2). Importantly, the combination of these three parameters outweighed the performance of each parameter taken separately to predict nasal high flow therapy outcome. Since its initial publication, several studies coming from different countries have confirmed the potential for the ROX index to predict need for intubation in patients with acute hypoxemic respiratory failure, thus making a valuable tool accessible to everyone, including nurses, to monitor on a routine basis. Because it reflects the patient's respiratory status, the greater the score, the better the patient's condition. Hence, one may hypothesize that, at the other end of the spectrum of respiratory failure (i.e., at the stage of weaning and withdrawal of the high flow device when the patient has considerably improved), the ROX index may also help identify those patients who will be successfully separated from the nasal high flow support. To date, one study has suggested that among several parameters, the value of the ROX index could be associated with successful cessation of nasal high flow. Here, in a retrospective exploratory study, investigators aim to to identify a cut-off value of the ROX index predictive of success of the withdrawal trial, to describe a one-year use of the withdrawal trial (average duration of use of nasal high flow before weaning, number of weaning trials, number of failed and successful weaning trials.); to describe the ROX value closest to weaning from nasal high flow, and to identify factors associated with success or failure of the withdrawal trial from nasal high flow therapy in patients receiving nasal high flow therapy; A successful withdrawal is defined as the withdrawal of nasal high flow without necessity of placing the patient back on nasal high flow within the following 24h. A failed withdrawal is defined by the need to resume nasal high flow within the 24h hours following the withdrawal. The possible identification of a cut-off value may help clinicians initiate earlier weaning from nasal high flow.

ELIGIBILITY:
Inclusion Criteria:

- ICU patient treated with nasal high flow

Exclusion Criteria:

* age < 18 years
* concomitant treatment with non-invasive ventilation
* acute hypercapnic respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients treated with nasal high flow therapy
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Value of the Respiratory Oxygenation index (ROX) at nasal high flow withdrawal | through each nasal high flow therapy, that lasts an average of 24hours
  the ROX index the closest to the time at which nasal high flow is withdrawn will be recorded

SECONDARY OUTCOMES:
use of nasal high flow before weaning | through each nasal high flow therapy, that lasts an average of 24 hours
  average duration of nasal high flow therapy before initiating a withdrawal trial (in hours)
number of withdrawal trials | through each nasal high flow therapy, that lasts an average of 24 hours
  the number of trials each patient will have performed will be recorded
number of patients who failed a withdrawal trial | throughout study duration which is a one-year period
  withdrawal failure is defined by patients who required to be placed back on nasal high flow after withdrawal of the high flow device within 24 hours of withdrawal.
number of patients who succeeded a withdrawal trial | throughout study duration which is a one-year period
  withdrawal success is defined by patients that have not required to be placed back on nasal high flow after withdrawal of the high flow device within 24 hours of withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Louis Mourier, Assistance Publique - Hôpitaux de Paris, Colombes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricard JD, Roca O, Lemiale V, Corley A, Braunlich J, Jones P, Kang BJ, Lellouche F, Nava S, Rittayamai N, Spoletini G, Jaber S, Hernandez G. Use of nasal high flow oxygen during acute respiratory failure. Intensive Care Med. 2020 Dec;46(12):2238-2247. doi: 10.1007/s00134-020-06228-7. Epub 2020 Sep 8. PMID 32901374
- [Background] Roca O, Caralt B, Messika J, Samper M, Sztrymf B, Hernandez G, Garcia-de-Acilu M, Frat JP, Masclans JR, Ricard JD. An Index Combining Respiratory Rate and Oxygenation to Predict Outcome of Nasal High-Flow Therapy. Am J Respir Crit Care Med. 2019 Jun 1;199(11):1368-1376. doi: 10.1164/rccm.201803-0589OC. PMID 30576221
- [Result] Rodriguez M, Thille AW, Boissier F, Veinstein A, Chatellier D, Robert R, Le Pape S, Frat JP, Coudroy R. Predictors of successful separation from high-flow nasal oxygen therapy in patients with acute respiratory failure: a retrospective monocenter study. Ann Intensive Care. 2019 Sep 11;9(1):101. doi: 10.1186/s13613-019-0578-8. PMID 31511996